CLINICAL TRIAL: NCT07303127
Title: Combination Effect of Bitter Melon (Momordica Charantia L.) Extract With Snakehead Fish (Channa Striata) Powder to Reduce the Glycaemia Increase in Type 2 Diabetes Mellitus
Brief Title: Combination of Bitter Melon Extract and Snakehead Fish Powder to Reduce Glycaemia in Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Muhammadiyah Surakarta (Other)
Responsible Party: Principal Investigator, Fahrun Nur Rosyid, Head of Quality Assurance Group, Universitas Muhammadiyah Surakarta
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMS-MOMORDICA-RCT2025
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
Keywords: AGEs; Bitter melon; Channa striata; Type 2 Diabetes Mellitus; Hypoglycaemic effect
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — bitter melon extract

STUDY DESIGN:
Intervention Model Description: A quasi-experimental parallel-group study in which participants are assigned to either the herbal supplement group or the placebo control group without randomization
Masking Description: Not applicable. This study did not implement masking; both investigators and participants were aware of group assignments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants in this arm receive a combination supplement containing bitter melon (Momordica charantia L.) extract and snakehead fish (Channa striata) powder. The supplement is administered in capsule form for 4 weeks in addition to their routine metformin therapy.
  Interventions: Dietary Supplement: Bitter Melon Extract and Snakehead Fish Powder Combination
- Control group (Placebo Comparator): Participants in this arm receive placebo capsules designed to match the appearance of the herbal supplement. The placebo is administered for 4 weeks while participants continue their routine metformin therapy.
  Interventions: Other: Placebo Capsule

INTERVENTIONS:
Dietary Supplement: Bitter Melon Extract and Snakehead Fish Powder Combination — Participants in the intervention group receive a combined herbal supplement consisting of bitter melon (Momordica charantia L.) extract and snakehead fish (Channa striata) powder. The supplement is prepared in capsule form at the Clinical Pharmacy Laboratory of Universitas Muhammadiyah Surakarta. Participants take the supplement daily for 4 weeks while continuing their routine metformin therapy. The formulation is standardized by maceration of bitter melon with ethanol followed by evaporation, and preparation of snakehead fish powder through steaming, drying, and milling before encapsulation.
  Arms: Intervention group
Other: Placebo Capsule — Participants in the control group receive placebo capsules that are visually identical to the herbal supplement capsules. The placebo contains inert, non-active ingredients and is administered daily for 4 weeks. The placebo is designed to match the appearance and dosing schedule of the active supplement but contains no bitter melon extract or snakehead fish powder. Participants continue their routine metformin therapy during the study.
  Arms: Control group

SUMMARY:
Type 2 Diabetes Mellitus (T2DM) is a chronic metabolic disorder characterized by persistent hyperglycemia, which contributes to the formation of advanced glycation end-products (AGEs) and increases the risk of long-term complications. Bitter melon (Momordica charantia L.) contains bioactive compounds that may support glycemic control, while snakehead fish (Channa striata) provides amino acids and fatty acids with potential antioxidant and restorative properties.

This study aims to evaluate the effect of a combined supplementation of bitter melon extract and snakehead fish powder on glycemic parameters in adults with T2DM. The study uses a quasi-experimental design with a control group, involving 80 participants recruited from community health centers in Surakarta, Indonesia. Participants are allocated to either a treatment group receiving the herbal combination or a control group receiving a placebo for four weeks.

Glycemic and biochemical parameters-including fasting plasma glucose, glycated albumin, insulin levels, and AGEs-are measured at baseline and at the end of the intervention period. Safety monitoring and adherence assessment are conducted throughout the study. This pilot investigation aims to explore the potential role of the combined supplement in the management of T2DM.

DETAILED DESCRIPTION:
Type 2 Diabetes Mellitus (T2DM) is a chronic metabolic condition marked by persistent hyperglycemia and associated inflammation, which contribute to the development of vascular and metabolic complications. Chronic hyperglycemia accelerates the formation of advanced glycation end-products (AGEs), which may impair tissue structure and function through oxidative stress and protein cross-linking mechanisms. Dietary phytochemicals and bioactive compounds have been increasingly studied as supportive strategies for glycemic regulation.

Bitter melon (Momordica charantia L.) has been traditionally used in various cultures as a natural remedy for diabetes. It contains several bioactive molecules, including alkaloids, flavonoids, catechins, saponins, charantins, and polypeptide-p, which are believed to contribute to glycemic regulation through mechanisms such as insulin secretagogue effects, enhancement of glucose utilization, modulation of glucose transporters, and inhibition of α-glucosidase activity. Despite its widespread traditional use, clinical findings have been variable due to differences in formulations, study durations, and methodological designs.

Snakehead fish (Channa striata) contains essential amino acids, fatty acids, and antioxidant components that may support metabolic processes and physiological recovery. While research has explored its nutritional and antioxidant potential, its combined use with bitter melon in T2DM has not been previously studied.

This study adopts a quasi-experimental design with a control group to assess the effect of a combined herbal supplement consisting of bitter melon extract and snakehead fish powder in individuals with T2DM. A total of 80 participants aged 25-65 years are recruited from four community health centers in Surakarta, Indonesia. Eligible participants have been clinically diagnosed with T2DM, are receiving metformin therapy, and meet specified biochemical inclusion criteria. Individuals with impaired renal or hepatic function, pregnancy, lactation, or known allergies to the study materials are excluded.

Participants provide informed consent and undergo initial screening before being allocated to either the treatment group or the placebo group. The intervention is administered for a period of four weeks. Outcome assessments include fasting plasma glucose, glycated albumin, insulin, and AGEs, measured at baseline and at the end of week four. Laboratory analyses utilize enzymatic methods and ELISA techniques. Medication adherence is monitored through pill counts and structured interviews during follow-up visits.

Throughout the study, participants are monitored for safety, tolerability, and any potential adverse events. This pilot study is intended to generate preliminary evidence on the feasibility and potential physiological effects of combining bitter melon extract and snakehead fish powder in the management of T2DM, and to inform the design of larger future clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Type 2 Diabetes Mellitus (T2DM).
* Age 25-65 years.
* Currently treated with one type of biguanide (metformin).
* Fasting plasma glucose 126-200 mg/dL.
* Willing to participate and sign informed consent.
* Able to attend all study visits at participating health centers.

Exclusion Criteria:

* Positive pregnancy test or currently breastfeeding.
* Impaired renal function (creatinine > 1.5 mg/dL).
* Impaired liver function (SGOT > 40 U/L or SGPT > 35 U/L, or ≥2× upper normal limit).
* Known allergy to bitter melon extract or snakehead fish powder.
* Any condition judged by investigators to interfere with study participation.
* Participants who withdraw consent or are unable to complete the intervention.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Fasting Plasma Glucose Level | Baseline and Week 4
  Fasting plasma glucose level measured using an enzymatic method to assess changes in glycemic status after 4 weeks of supplementation. Blood samples are collected after an overnight fast at baseline and at the end of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Faculty of Health Sciences FIK UMS, Principal Investigator — Universitas Muhammadiyah Surakarta
Locations (1):
- Faculty of Health Sciences, Universitas Muhammadiyah Surakarta, Surakarta, Centre Java, Indonesia

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the study was conducted as a small pilot trial with limited sample size, and the informed consent obtained from participants did not include permission for public or external data sharing. Additionally, privacy protections and institutional policies restrict the distribution of raw participant-level data outside the research team.